CLINICAL TRIAL: NCT00258063
Title: Open-Label, Randomized, Partially Balanced, Incomplete Block Design Study to Evaluate the Hormone Exposure From Commercial EVRA (Manufactured by LOHMANN Therapie-Systeme) and an Oral Contraceptive
Brief Title: A Study to Evaluate the Exposure of Norelgestromin and Ethinyl Estradiol From Commercial Lots of EVRA (a Transdermal Contraceptive Patch Manufactured by LOHMANN Therapie-Systeme) and CILEST (an Oral Contraceptive)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR002212
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Contraception; Female Contraception
Keywords: Transdermal contraception; contraceptive; hormonal, steroid contraception; ethinyl estradiol; progesterone; EVRA; CILEST; ORTHO EVRA
MeSH Terms: interventions — norelgestromin; Ethinyl Estradiol

INTERVENTIONS:
Drug: EVRA® transdermal contraceptive patch containing 6 mg of norelgestromin and 0.60 mg of ethinyl estradiol (versus CILEST® tablets).

SUMMARY:
The objective of this study is to estimate exposure to the hormones norelgestromin, norgestrel, and ethinyl estradiol in healthy female volunteers across multiple commercial lots of EVRAÂ® (a transdermal contraceptive patch manufactured by LOHMANN Therapie-Systeme), to compare these data to exposure data from one clinical lot, and to compare these data to exposure data from a commercially available oral contraceptive.

DETAILED DESCRIPTION:
This single-center, open-label, randomized, partially-balanced, incomplete block design study will consist of a pre-treatment phase (a screening period lasting up to 21 days), an open-label treatment phase (three 7-day treatment periods separated by 21-day washouts), and a post-treatment phase (a follow-up or early withdrawal visit). Total participation in the study is approximately 67 days. Approximately 54 subjects will be enrolled. The study population comprises healthy women, ages 18 to 45 years inclusive, who weigh at least 110 pounds, have a body mass index (BMI) between 16 and 29.9 kg per meter squared.

Subjects will wear an EVRA® patch or take CILEST® during each of the three 7-day treatment periods; treatment periods will be separated by a 21-day washout period. When a subject is to wear EVRA®, a patch from 1 of the 6 selected commercial lots will be applied on the buttock and worn for 7 days. Patches will be applied by the investigator or designated study unit personnel. All patches will be worn on the upper outer quadrant of the same buttock, but not necessarily in the exact same position. The investigator or designated study unit personnel will remove the patches and will evaluate the adhesion of the patches before removal. When a subject is to receive CILEST®, tablets from 1 of the 3 selected commercial lots will be administered daily for 7 consecutive days. A minimum of 21 days after removal of the patch or the seventh dose of CILEST®, the subject will begin another treatment period, until she completes 3 open-label treatment periods.

Subjects will be confined to the study unit for blood sample collections for determination of NGMN, NG, and EE plasma concentrations. Blood samples will be collected (via venipuncture) immediately before each dose and at specified time points after each dose is administered. Pharmacokinetic parameters of NGMN, NG, and EE, including Cmax, tmax, and AUC, after each treatment will be estimated by standard methods. Safety will be assessed throughout the study, and will be based on adverse events and changes in physical and gynecologic examinations (including breast examinations), vital signs, electrocardiograms (ECGs), and clinical laboratory test results. Three 7-day treatment periods; treatments separated by 21-day washout. Based on the randomization schedule, some subjects will wear an EVRA® patch in all 3 periods (on the upper outer quadrant of the buttock for 7 days), some will wear a patch in 2 periods and take CILEST® oral tablets once daily in 1 period, and some will wear a patch in 1 period and take CILEST® oral tablets once daily in 2 periods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are not pregnant (as demonstrated by negative pregnancy tests at screening and before admission for each treatment period) and who have completed their last term pregnancy at least 60 days before the admission visit
* confirmed to be in good health as determined by medical history, physical examination (including vital signs), gynecologic examination (including breast examination), and laboratory test results
* have a history of regular menstrual cycles, weigh at least 110 pounds (50 kilograms), have a body mass index (BMI) between 16 and 29.9 kg per meter squared, a hematocrit of at least 36% at screening, and a ferritin level above the lower limit of normal
* are nonsmokers and have not used any tobacco products for at least 6 months before study admission
* agree not to use any prescription or nonprescription medications for the duration of the study, and if the subject or her male partner are not surgically sterile, agree to continue to use a non-hormone-containing intrauterine device (IUD) or one of the following methods of double-barrier contraception during participation in the study: condoms and foam, diaphragm and gel, or cervical cap and gel.

Exclusion Criteria:

* Subjects with a history or presence of disorders commonly accepted as contraindications to sex hormonal therapy including, but not limited to: deep vein thrombophlebitis or thromboembolic disorders, cerebral vascular or coronary artery disease, chronic untreated hypertension or migraines, benign or malignant liver tumor which developed during the use of oral contraceptives or other estrogen-containing products, or known or suspected estrogen-dependent neoplasia
* presence of disorders commonly accepted as contraindications to combined oral contraceptive therapy including, but not limited to: undiagnosed abnormal vaginal bleeding, any neurovascular lesion of the eye or serious visual disturbance, any impairment of liver function, liver disease, or kidney disease
* currently pregnant or breast feeding, or have evidence of cervical dysplasia (as documented by a Pap smear within 6 months before randomization)
* has used steroid hormonal therapy within 30 days before the first admission visit, received a Depo Provera® injection within 6 months of the first admission visit, received a Lunelle® injection within 60 days before the first admission visit, currently has Norplant® in place, or has had removal of Norplant within the 60 days before the first admission visit, or has used a steroid hormone-containing intrauterine device (IUD) within 3 months of randomization
* has elevated blood pressure (sitting systolic BP >140 mm Hg and/or diastolic BP >90 mm Hg)
* has a history or presence of hypersensitivity in response to topical applications (bandages, surgical tape, etc.) or has active inflammation of the skin (dermatitis) or other skin conditions (dermatosis).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-05; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
A comparison of exposure and pharmacokinetics for norelgestromin, (NGMN), norgestrel (NG), and ethinyl estradiol (EE) for EVRA®, CILEST® and historical data from one ORTHO EVRA® clinical development lot.

SECONDARY OUTCOMES:
An assessment of safety from screening to final visit (incidence of adverse events, changes in physical, gynecologic and breast examinations, vital signs, laboratory tests and electrocardiogram results).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Open Label, Randomized, Partially Balanced, Incomplete Block Design Study to Evaluate the Hormone Exposure From Commercial EVRA� Manufactured by LOHMANN Therapie Systeme and an Oral Contraceptive — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=458&filename=CR002212_CSR.pdf